CLINICAL TRIAL: NCT03789058
Title: Efficacy of Non-Steroidal Anti-Inflammatory Drug (Ibuprofen) Chronotherapy in Healing After Surgical Extraction of the Mandibular Third Molar - A Randomized Clinical Trial Protocol
Brief Title: Efficacy of Ibuprofen Chronotherapy in Healing After Surgical Extraction of the Mandibular Third Molar
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: McGill University (Other); InterPharma One LLC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20170307
Record Dates: First submitted 2018-12-23; First posted 2018-12-28 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Operation Site Inflammation; Pain, Postoperative; Teeth, Impacted
MeSH Terms: conditions — Pain, Postoperative; Tooth, Impacted | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment a single-center double-blind randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: The treatment regimens were masked for both participants and care provider (Clinical investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical with conventional NSAID 3 times/day (Active Comparator): Control group will have surgical intervention to remove wisdom tooth and receive conventional NSAID treatment three times per day
  Interventions: Drug: Ibuprofen 400 mg
- Surgical with conventional NSAID 2 times/days (Experimental): The experimental group will have surgival intervention to remove wisdom tooth and receive NSAID treatment only two times per day: once after breakfast and once after lunch, but not at night.
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Surgical removal of wisdom teethb with different regimen of Ibuprofen frequency ; three times versus two times .
  Other Names: Advil; Motrin

SUMMARY:
Clinical and preclinical studies have demonstrated encouraging results of non-steroidal anti-inflammatory drug (NSAID) chronotherapy in the management and treatment of inflammatory diseases such as rheumatoid arthritis. However, no previous clinical trials have addressed how the timing of NSAID administration within the day affects pain and healing outcomes after oral surgery that involves bone removal, such as surgical extraction of the third molars. Methods to address our aim, Single-center double-blind randomized controlled trial study design has been adopted. Patients who needed a lower third molar extraction and meet the eligibility criteria will be recruited. Participants will be randomized into two groups. Subjects in group one will be instructed to take an NSAID (ibuprofen 400 mg) at 7 AM and 12 PM combined with a placebo before bed between 8 and 10 PM for three days postoperatively. Subjects in group 2 will be instructed to take an NSAID (ibuprofen 400 mg) between 7 AM, 12 PM and between 8 and 10 PM for three days postoperatively. The patients' self-reported pain in the three days after surgery will be recorded as the primary outcome.

Additionally, healing indicators such as the maximum interincisal distance and measurements of facial swelling will be recorded preoperatively and four days postoperatively. Each participant's blood level of C-reactive protein will be recorded pre- and postoperatively as an inflammatory marker.

Discussion:

The study will estimate the effect of using NSAID only in the morning following surgical extraction of the third molar to decrease pain and improve postoperative healing and recovery in comparison to the routine use of NSAIDs three times per day.

DETAILED DESCRIPTION:
Introduction and background:

The surgical extraction of wisdom teeth under local anesthesia is one of the most common oral surgical procedures (1). Ten million third molars (wisdom teeth) are extracted from approximately 5 million people in the United States of America each year at an annual cost of over $3 billion. Additionally, more than 11 million patient-days of "standard discomfort or disability" were reported due to surgical removal of wisdom teeth, with an average of 4.9 lost work days per procedure (2, 3). Most of wisdom teeth surgical extractions require bone removal (4). Bone removal is associated with a broad range of postoperative discomfort and complications (e.g., pain, swelling, bruising, and malaise). Most of these complications are initiated by the inflammatory process from traumatic injury to the bone during the surgery. Currently, postoperative pain management is limited to acetaminophen, opioids and NSAIDs (5, 6). However, these drugs are all problematics. Acetaminophen is not effective in managing severe pain (6). Opioids and NSAID are effective in pain management, but opioids can cause constipation and addiction (7, 8), While NSAIDs may delay bone healing (9, 10). Dentists and maxillofacial surgeons all over the world prefer to prescribe NSAID after this type of surgery (11). The mechanism of action of NSAIDs is the reversible inhibition of the enzyme cyclooxygenase (COX), which is believed to be responsible for the synthesis of prostaglandins (PGs) (10). Prostaglandins play a major role in inflammatory and nociceptive processes (12). Two isoforms of COX, namely, COX-1 and COX-2, are responsible for the synthesis of PG from arachidonic acid (AA). Both have essential roles in the inflammatory process after bone surgery, but COX-1 is involved more in the integrity of the gastrointestinal tract and renal tract tissue, while COX-2 is mainly involved in the inflammatory and healing process later (13). NSAIDs are either nonselective (inhibiting both COX-1 and COX-2) or selective (inhibiting COX-2 only). Ibuprofen is a peripherally acting analgesic with potent anti-inflammatory action that works through reversible and balanced COX-1/ COX-2 inhibition, which provides faster and more effective analgesia than many other NSAIDs without any apparent increased safety risk (14). Ibuprofen is routinely used in the treatment of moderate to severe acute pain in the general population, including dantal pain (15-17). Results from Cochrane systematic reviews demonstrate that higher doses and frequencies of NSAID use are associated with better pain control after dental (wisdom tooth extraction) and non-dental surgeries (9, 18, 19). Increasing the dose and frequency of NSAIDs was associated with an increased risk of adverse effects. Despite the promising results associated with the use of different NSAIDs for pain control after wisdom tooth surgeries, patients still report pain and other discomfort indicators such as swelling and trismus, especially during the first three days after the procedure (20). These symptoms can affect patient's life, including activities of daily living and even quality of life (3, 20-22). Animal studies suggest that NSAID affect bone healing outcomes such as biomechanical measuments and number of bones with non-unions (23-35). Some authors have even compared the effect of NSAIDs on fracture healing with those of other pharmacological agents such as steroids (36, 37). Høgevold et al, demonstrated that short-term administration of some anti-inflammatories, such as indomethacin, inhibits fracture healing, while methylprednisolone does not (36). Bhattacharyya et al. reported that patients receiving NSAIDs within 90 days after fracture had a 3.7-fold risk of nonunion, while the risk for opioid users was 1.6-fold (38). Clinical trials in humans pose some challenges, especially the need to control confounders such as smoking, diabetes, obesity and other factors that are associated with the healing of long-bone fractures (6, 39). Four retrospective studies suggested that patients using NSAIDs after fracture had a higher incidence of non-union compared to those that did not use NSAIDs (38, 40-42). All living organisms possess a circadian rhythm that anticipates the response to changes during the 24-hour cycle (43). The circadian system in mammals is composed of a central clock within the suprachiasmatic nuclei and a peripheral clock inside all cells. The circadian clock is controlled through a feedback loop featuring a heterodimer of two core clock gene products: circadian locomotor output cycles kaput (Clock) and brain and muscle Arnt-like protein-1 (Bmal1). Clock and Bmal1 drive the expression of two inhibitors, cryptochrome (Cry) and period (Per) (44). This molecular clock modulates the immune response and bone healing process (44). The circadian rhythms in the expression of various cytokines by immune cells are presented in Table S1. Macrophage activity, leukocyte recruitment, and proinflammtory mediators such as interleukin-1β (IL-1β), IL-6, and IL-12 increased at the beginning of the daily activity phase.

During the active phase, there are also increased levels of Toll-like receptors TLR9 and TLR4, which upregulate the expression of CCL2, CXCL1, and CCL5, leading to leukocyte recruitment and potential tissue damage at the injured site (43-46)(Fig.1.). On the other hand, anti-inflammatory mediators and other growth and angiogenesis factors, such as vascular endothelial growth factor (VEGF), peak during the resting phase (44, 47, 48) (Table S2.). The 24-hour circadian rhythm oscillation occur in bone tissue during growth (49), formation, resorption (50, 51), and endochondral ossification during fracture bone healing (51). Experimental studies in rodents and humans reveal that disruption of sleep and circadian rhythm impair bone formation (52). All bone cells such as osteoblasts, osteoclasts, and chondrocytes express clock genes that influence bone volume regulation, such as Per or Cry (53, 54). The circadian clock also affects pain, with sensitivity peaking during the active phase (55). Part of the pain response oscillation could be explained by changes in COX-1 and COX-2 activity throughout the day (56), especially after an injury or insult (57). These variations may contribute to the clinical evidence of circadian and circannual variations in the pharmacokinetics effects of NSAID. Specifically, maximum absorption and effectiveness are achieved when the drug is administered during the active phase (58-62). We performed experimental studies to estimate the extent to which the timing of NSAID doses can affect animal pain behaviour and recovery after bone fracture surgery. We used a validated model of fracture healing in young female mice. The results showed that administration of NSAIDs during the active phase after tibia fracture surgery, compared to administration during the resting phase, significantly attenuated the pain response and improved the mechanical and histomorphometric properties of the healing callus. Recent evidence suggests that the timing of skin wounds or surgery affects healing and postoperative recovery after cardiovascular surgeries (63, 64). The chronotherapeutic use of anti-inflammatory medications after oral surgeries is of clinical importance, especially with increasing evidence regarding the clinical efficacy of this approach in medicine. No clinical studies have investigated the effectiveness of this approach after minor oral surgeries. Expected contribution and research question The overarching aim of this study is to contribute evidence regarding the efficacy of NSAID chronotherapy in patient recovery from wisdom tooth surgery. This is an important aim considering that the outcomes of this investigation can be used for other medical interventions involving bone healing. The research question is as follows: among patients undergoing surgical extraction of wisdom teeth, to what extent does a morning doses of ibuprofen 400 mg, in comparison to a routine dose schedule of three times per day, decrease patients' pain and improve wound healing when taken for three days after surgery .

ELIGIBILITY:
Inclusion Criteria:

(i) be aged between 18 and 35 years old

(ii) be healthy according to the American Society of Anesthesiologists (ASA) classification (subject should not have an active infection, trismus, hyperthermia, or swelling before surgery and must be able to maintain adequate oral hygiene)

(iii) have an adequate understanding of written and spoken English or Arabic to fill out a questionnaire,

(iv) be capable of signing an informed consent form

(vi) third molar surgical extraction, the indicated teeth should be lower third molars and partially or completely impacted

Exclusion Criteria:

(i) have a history of systemic diseases (e.g., diabetes mellitus, hypertension, gastric ulcer)

(ii) have a severe/serious illness that requires frequent hospitalization

(iii) are current smokers

(iv) are pregnant or breastfeeding

(v) are taking antinflammtory or analgesic drugs in the previous two weeks or are allergic to NSAIDs

(vi) have impaired cognitive or motor function

(vii) are unable to return for evaluations/study recalls.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain Measurement | four days measurement of VAS
  Measuring of post operative pain severity according to Visual Analogue Scale healing indicators such as edema and mouth opening .

SECONDARY OUTCOMES:
Inflammation Degree Measurement | Pre-Op, 4th day after operation
  Inflammation Degree by measuring C-reactive Protein (CRP)
Facial Swelling and mouth opening measuring | pre-op, 4th day post op.
  Facial Swelling will be measured according to LASKIN method

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Z Tamimi, HSD, Principal Investigator — JUST
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
data will be provided upon request or required for publication .